CLINICAL TRIAL: NCT01790568
Title: Pilot Trial of Vorinostat Plus Tacrolimus & Methotrexate to Prevent Graft Versus Host Disease Following Unrelated Donor Allogeneic Transplant
Brief Title: Vorinostat Plus Tacrolimus & Methotrexate to Prevent Graft vs Host Disease Following Unrelated Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UMCC 2012.047; HUM00070080 (Other: University of Michigan)
Record Dates: First submitted 2012-10-02; First posted 2013-02-13 (Estimated); Results first posted 2018-01-02 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-07

CONDITIONS: Graft vs Host Disease; Hematologic Neoplasms; Non-Neoplastic Hematologic and Lymphocytic Disorder
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms | interventions — Vorinostat; Tacrolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat (Experimental): Vorinostat, in combination with standard of care medications tacrolimus and methotrexate, for GVHD prophylaxis after unrelated donor stem cell transplant.
  Interventions: Drug: Vorinostat; Drug: Tacrolimus; Drug: Methotrexate

INTERVENTIONS:
Drug: Vorinostat — administered at a dose of 100 mg orally, twice daily starting on day -10 in order to achieve steady-state prior to beginning the conditioning chemotherapy, and continued after transplant (day 0) until day +100.
  Other Names: Zolinza
Drug: Tacrolimus
Drug: Methotrexate

SUMMARY:
This protocol, UMCC 2012.047, was a pilot study initially intended for 12 subjects. After completing enrollment of the planned 12 subjects, we are extending the study to an additional 25 subjects. The trial will examine the safety and efficacy of the addition of vorinostat, the study drug, to standard medications to try to prevent or lower the risk of graft versus-host disease (GVHD) for recipients of unrelated (matched) donor, blood or marrow stem cell transplants. The transplant regimens, chosen according to current institutional policy, will depend upon the recipients underlying disease (their blood cancer or other blood disorder), previous therapy, and current health issues. GVHD prophylaxis (preventive drug intervention) will be the local institutional standard for post-transplant immunosuppression, including tacrolimus and methotrexate, plus vorinostat. Vorinostat will be given twice daily orally beginning 10 days prior to the recipient's transplant and continue for up to 100 days after transplant.

DETAILED DESCRIPTION:
This trial is investigating the use of vorinostat (Merck) for standard graft versus-host disease (GVHD) prophylaxis after unrelated donor allogeneic hematopoietic cell transplantation (HCT). A major limitation of the increased utilization of allogeneic HCT (Hematopoietic Cell Transplantation) is the inferior outcomes when donors other than HLA (HumanLeukocyte Antigen)-matched siblings are used. Compared to matched related donors, recipients of matched unrelated donor transplants are at a significantly increased risk of death and transplant-related mortality (TRM). Acute GVHD remains a significant contributor to TRM, which develops in approximately 50-70% of recipients receiving these type of grafts despite standard immunosuppressive prophylaxis. Thus, novel GVHD prophylaxis strategies which successfully attenuate acute GVHD-related complications without increasing other causes of TRM or relapse are needed.

The historical experience of day 100 grade 2-4 acute GVHD in 154 comparable patients treated at the University of Michigan (2005 - 2011) receiving standard GVHD prophylaxis after unrelated donor allogeneic transplant is 48%. At Washington University, the cumulative incidence of acute grade 2-4 GVHD in patients following unrelated donor transplant is 62%.

Research data collectively suggests, that reducing lethal acute GVHD should improve long-term survival for patients undergoing unrelated donor transplant.

ELIGIBILITY:
Inclusion Criteria:

* A prospective patient for allogeneic HSCT for hematologic conditions, both malignant and non-malignant. Donor can be unrelated marrow or peripheral blood cells. A patient with history of CNS involvement is eligible if CNS disease is in remission at time of study consideration.
* Age between 18-75 years
* The donor and recipient must have an HLA-8/8 allelic match at the HLA-A, -B, -C, and -DRB1.
* Diagnosis of following diseases (subject to additional complex screening criteria)

  * Acute Myelogenous Leukemia:

    * First remission (cytogenetic intermediate or high risk)
    * Second or subsequent remission
  * Chronic Myelogenous Leukemia:

    * First, subsequent chronic phases, or atypical
    * Accelerated Phase
  * Myelodysplastic syndromes
  * Chronic Lymphocytic Leukemia
  * Primary Myelofibrosis
  * Mature B Cell Malignancies (including Mantle Cell Lymphoma, Follicular Lymphoma. Diffuse Large B Cell Lymphoma, Non-Hodgkin Lymphoma not otherwise specified)
* Karnofsky (Attempt to classify a cancer patients' activities of daily life that runs from 0 to 100 where 100 represents perfect health and 0 represents death) >70%
* Life expectancy of greater than 6 months.
* Organ and marrow function as defined by the institutional BMT (Bone Marrow Transplant) program clinical practice guidelines
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Able to swallow capsules/tablets

Exclusion Criteria:

* Not a candidate for an unrelated donor allogeneic transplant conditioning regimen based on the current institutional BMT program clinical practice guidelines. Organ function criteria will be utilized per the current institutional BMT program clinical practice guidelines. There will be no restriction to study entry based on hematological parameters.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat
* Undergoing a total body irradiation (TBI)-based conditioning regimen (TBI 1200 cGy)
* Uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Patients still under therapy for presumed or proven infection are eligible provided there is clear evidence (radiographic findings and/or culture results) that the infection is well-controlled. Patients under treatment for infection will be enrolled only after clearance from the PI
* Any medical or psychological comorbidities/conditions that would keep the patient from complying with the needs of the protocol and/or would markedly increase the risk of morbidity and mortality.
* Pregnant women or nursing mothers.
* Evidence of HIV seropositivity and/or positive PCR assay, HTLV1 / HTLV2 seropositivity.
* Evidence of Hepatitis B or Hepatitis C PCR positivity.
* Less than 18 years of age.
* A history of prolonged QTc syndrome.
* Taking or have had prior treatment with a drug like vorinostat within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-12; Primary Completion 2017-01-01 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pavan Reddy, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Choi SW, Braun T, Henig I, Gatza E, Magenau J, Parkin B, Pawarode A, Riwes M, Yanik G, Dinarello CA, Reddy P. Vorinostat plus tacrolimus/methotrexate to prevent GVHD after myeloablative conditioning, unrelated donor HCT. Blood. 2017 Oct 12;130(15):1760-1767. doi: 10.1182/blood-2017-06-790469. Epub 2017 Aug 7. PMID 28784598

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 patients were enrolled in the initial NCI funded portion of the Vorinostat trial (NCT1789255). 26 were enrolled to the expansion of that trial (NCT01790568). 1 pt removed prior to transplant so 25 were evaluable. All patients were treated identically. Although 26 patients were enrolled to this portion of the trial, ALL 37 are analyzed together.
Groups:
- Vorinostat: NCI sponsored pilot trial of Vorinostat, in combination with standard of care medications tacrolimus and methotrexate, for GVHD prophylaxis after unrelated donor stem cell transplant.
  Vorinostat: administered at a dose of 100 mg orally, twice daily starting on day -10 in order to achieve steady-state prior to beginning the conditioning chemotherapy, and continued after transplant (day 0) until day +100.
- Vorinostat Expansion: Expansion of the NCI sponsored pilot trial of Vorinostat, in combination with standard of care medications tacrolimus and methotrexate, for GVHD prophylaxis after unrelated donor stem cell transplant.
  Vorinostat: administered at a dose of 100 mg orally, twice daily starting on day -10 in order to achieve steady-state prior to beginning the conditioning chemotherapy, and continued after transplant (day 0) until day +100.
Period: Overall Study
Arm/Group | Vorinostat | Vorinostat Expansion
Started | 12 | 26
Completed | 12 | 25
Not Completed | 0 | 1
Not completed — Progression prior to transplant | 0 | 1

BASELINE CHARACTERISTICS:
Population: This trial consisted of an initial pilot phase, funded by the NCI, that enrolled 12 patients (NCT01789255). The trial was extended to enroll an additional 25 patients. The results presented here include information for all 37 patients.
Arm/Group | Vorinostat
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 56 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White, non-hispanic | 33
  Race/Ethnicity: White, Hispanic | 2
  Race/Ethnicity: Asian | 1
  Race/Ethnicity: Not reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients That Experience Grade 2-4 GVHD Within 100 Days of Transplant
Description: GVHD Staging:
  Grade 2: (Skin) Maculopapular rash 25-50% BSA, (Liver) bilirubin 3.1-6mg/dl, (Gut) 1000-1500 ml/day for adult and 20-30ml/kg/day for child.
  Grade 3: (Skin) Maculopapular rash >50% BSA, (Liver) 6.1-15mg/dl, (Gut) >1500mg/day for adult and >30ml/kg/day for child.
  Grade 4: (Skin) Generalized erythroderma plus bullous formation and desquamation >5% BSA, (Liver) >15mg/dl, (Gut) Severe abdominal pain with or without ileus, or grossly bloody stool.
Time Frame: 100 Days
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vorinostat
Number analyzed (Participants) | 37
percentage of patients | 22 [11 to 39]

2. Secondary Outcome: Percentage of Patients Alive at 1 Year
Description: Overall survival at 1 Year.
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vorinostat
Number analyzed (Participants) | 37
percentage of patients | 76 [63 to 92]

3. Secondary Outcome: Non-Relapse Mortality Incidence
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Vorinostat
Number analyzed (Participants) | 37
percentage of patients | 16 [7 to 34]

ADVERSE EVENTS:
Time Frame: Toxicity was assessed weekly through day +100 after transplant, then monthly through day +180.
Arm/Group | Vorinostat
All-Cause Mortality (participants affected / at risk) | 10/37
Serious Adverse Events (participants affected / at risk) | 24/37
Other Adverse Events (participants affected / at risk) | 26/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat (N=37)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 3 (3)
Immune system disorders - Other (Immune system disorders) | 6 (6)
Abdominal infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 4 (4)
Lung infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Radiculitis (Nervous system disorders) | 1 (1)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat (N=37)
anemia (Blood and lymphatic system disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 7 (12)
Vomiting (Gastrointestinal disorders) | 4 (7)
Pain (General disorders) | 1 (1)
Immune system disorders - Other (Immune system disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (3)
Creatinine increased (Investigations) | 6 (7)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (5)
Platelet count decreased (Investigations) | 13 (15)
White blood cell decreased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes